CLINICAL TRIAL: NCT01606605
Title: Retrospective Analysis of Diffuse Large B-cell Lymphoma: Identification of Factors Associated With Treatment Resistance Via Gene Expression Profile
Brief Title: Treatment Resistance Related With Gene Expression Profile of Diffuse Large B-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Other Study IDs: 2010-05-025
Record Dates: First submitted 2012-05-22; First posted 2012-05-25 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Lymphoma; Prognosis; Relapse; Gene; microRNA
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Parrafin-embedded tissue blocks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diffuse large B-cell lymphoma: Patients diagnosed and treated at the Samsung Medical Center

SUMMARY:
The investigators perform a retrospective microarray gene expression profiling study of FFPE from a cohort of DLBCL patients with whole genome cDNA mediated Annealing Selection and Ligation (WG-DASL) assay. The investigators also study the pattern of microRNA from patients with diffuse large B-cell lymphoma. The results of gene expression profiles and microRNA is correlated with clinical outcomes of diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
1. Whole genome cDNA mediated Annealing Selection and Ligation (WG-DASL) assay

   * Diffuse large B-cell lymphoma patients
   * Paraffin-embedded tissue
   * End points: Progression-free survival, overall survival
   * Statistics: Leave one-out method
2. Nano string assay for microRNA

   * Diffuse large B-cell lymphoma patients
   * Paraffin-embedded tissue
   * End points: Progression-free survival, overall survival
   * Statistics: Leave one-out method

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diffuse large B-cell lymphoma
* Patients with tissue blocks available for study
* Patients with adequate medical records

Exclusion Criteria:

* Patients diagnosed with other subtypes of lymphoma

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diffuse large B-cell lymphoma
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who relapse or progress after 1st line chemotherapy | two years

SECONDARY OUTCOMES:
Number and type of genes and microRNA which are significantly related with relapse or progression (P < 0.05) | two years

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Medical Center Cancer Research Institute
Locations (1):
- Samsung Cancer Research Institute, Seoul, South Korea